CLINICAL TRIAL: NCT06319885
Title: Text Messaging to Reduce High-risk Alcohol Use Among Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Anette Søgaard Nielsen, PhD (Unknown); Kjeld Andersen, PhD (Unknown); Angelina Mellentin, PhD (Unknown); Alexis Kuerbis (Unknown)
Responsible Party: Principal Investigator, Silke Behrendt, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SDU project nr. 3110386; ID: 158341 (Other Grant/Funding Number: Trygfonden)
Record Dates: First submitted 2024-03-04; First posted 2024-03-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Hazardous Alcohol Use
Keywords: older adults; digital intervention; prevention; text messaging

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either one out of six intervention conditions with different types of text messaging (including one assessment-only control condition).
Who Masked: Participant
Masking Description: Participants are informed in the study material that they are allocated to groups that receive different text messages. They receive no further information on the intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Gain-framed (Experimental): One daily text-message and weekly alcohol use assessment. The text-messages focus on the positive consequences of drinking less.
  Interventions: Behavioral: Text messaging
- Loss-framed (Experimental): One daily text-message and weekly alcohol use assessment. The text-messages focus on the negative consequences of a high alcohol-intake.
  Interventions: Behavioral: Text messaging
- Static-tailored (Experimental): One daily text-message and weekly alcohol use assessment. The text-messages are adapted to the participant's gender and to baseline information on (e.g.) participants' drinking patterns, social network, and self-efficacy. One message per week is adapted to the day on which the participants find it most challenging to reduce their drinking.
  Interventions: Behavioral: Text messaging
- Adaptive-tailored (Experimental): One daily text-message and weekly alcohol use assessment. The text-messages are adapted to the participant's gender and to baseline information on (e.g.) participants' drinking patterns, social network, and self-efficacy. One message per week is adapted to the day on which the participants find it most challenging to reduce their drinking. In addition, text messages are adapted to the weekly alcohol-assessment over time and participants can demand supportive Just-In-Time messages.
  Interventions: Behavioral: Text messaging
- Combined (Experimental): This arm combines all features of the arms Adaptive-tailored and Gain-framed.
  Interventions: Behavioral: Text messaging
- Assessment-only (No Intervention): The control group. Participants do only receive 4 questions on their alcohol intake once a week.

INTERVENTIONS:
Behavioral: Text messaging — Participants receive text messages related to their alcohol consumption.
  Arms: Adaptive-tailored; Combined; Gain-framed; Loss-framed; Static-tailored

SUMMARY:
High-risk drinking is very prevalent among Danes aged 55+. It poses a serious risk to health and independent living, burdening health care systems and family members. Measures to reduce high-risk alcohol use in this growing group at need are urgently needed. A recent small study from the US shows that text messaging reduces high-risk alcohol intake in older adults. The investigators will conduct a pilot study with the same intervention in Denmark, with adaptations to language and culture. The pilot study will investigate among Danish older adults whether text messaging is well-accepted by participants and feasible in terms of reducing 1) high-risk drinking and 2) commonly accompanying problems with daily functioning, social relationships, and mental and physical health. The pilot-trial will include n=60 adults aged 55-80 years who will receive alcohol-related text messages (within a secure app for data protection purposes) over 12 weeks. Assessments will include a baseline assessment and a post-assessment.

ELIGIBILITY:
Inclusion Criteria:

* consumption of > 10 standard drinks á 12 gram ethanol per week (i.e., high-risk alcohol use defined by the Danish Health Authority) in the past four weeks
* desire to reduce drinking
* age 55 to 80 years
* mobile phone ownership and willingness to receive and respond to text messages
* fluency in Danish.

Exclusion Criteria:

* drinking more than 53 standard drinks per week in the last four weeks
* past 12 month alcohol withdrawal symptoms or lifetime history of serious withdrawal symptoms (e.g., seizures)
* score above 12 on the Short alcohol withdrawal scale; SAWS
* possible drug dependence (i.e., use of illegal drugs or psychotropic medication taken without prescription more than once a month)
* indication of serious psychiatric illness (lifetime diagnosis of psychosis or bipolar disorder, inpatient treatment or medication for these, recent suicidality)
* current alcohol/drug abuse treatment or a desire to start alcohol/drug abuse treatment during the study
* medical condition that requires abstinence from alcohol
* wish to achieve abstinence (applied to secure a focus on reduction)
* lack of understanding of study protocol or reading difficulty as evidenced by a score of less than 7 out of 10 on the consent form quiz.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
High-risk alcohol use (yes/no) | Assessed at 12 weeks after baseline, alcohol use through the past seven days
  Drinking over 120 gram ethanol in seven days (determined by outcomes 4 & 5 )

SECONDARY OUTCOMES:
WHOQOL-Bref (The World Health Organization Quality of Life Brief Version ) | Assessed at 12 weeks after baseline
  Quality of life, functioning. Higher scores represent higher quality of life.
OBSESSIVE-COMPULSIVE DRINKING SCALE (OCDS) | Through the past seven days, assessed at 12 weeks after baseline
  Degree of compulsive alcohol use, with higher scores representing a higher degree
Drinker Inventory of Consequences (DrInC-2R) | Through the past 14 days, assessed at 12 weeks after baseline
  Consequences of drinking, a higher score represents greater consequences
Frequency of alcohol use | Assessed at 12 weeks after baseline, alcohol use through the past seven days
  Measured in number of days
Amount of alcohol use | Assessed at 12 weeks after baseline, alcohol use through the past seven days
  Measured in standard drinks with one drink equivalent to 12 gram pure ethanol
Heavy drinking days | Assessed at 12 weeks after baseline, alcohol use through the past seven days
  Count, number of days with 5 or more standard drinks
User evaluation (tailor-made) | Assessed at 12 weeks after baseline, through 12 weeks (the intervention period)
  Subjective evaluation of user-friendliness, quality of the messages, and cultural adaptation (participants rate the intervention on a scale from 0= do not agree at all through 6= fully agree). Participants also tick off boxes for simple questions on other help received in the study period and on their impressions of the language and cultural appropriateness.
PHQ-9 (Patient Health Questionnaire-9 ) | Assessed at 12 weeks after baseline, through the past 14 days
  A higher score represents a greater degree of depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Silke Behrendt, PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark, Department of Psychology, Odense, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No